CLINICAL TRIAL: NCT01351155
Title: Comparison of Three Devices to Prevent Skin Damage Induced by Facial Mask Ventilation During Acute Respiratory Failure: a Multicenter Randomised Controlled Study
Brief Title: Prevention of Damage Induced by Facial Mask Ventilation
Acronym: 3PROSNIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale San Donato (Other)
Collaborators: Smith & Nephew, Inc. (Industry); Italian Association of Hospital Pneumologists (Other)
Responsible Party: Principal Investigator, Raffaele Scala, MD, Ospedale San Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RSAIPO2011
Record Dates: First submitted 2011-05-05; First posted 2011-05-10 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Acute Respiratory Failure
Keywords: acute respiratory failure; noninvasive ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- polyurethane foam (Allewyn adesive) (Active Comparator): Polyurethane foam is applied as skin protective dressing device before NIV and kept on site till the 7th day of treatment Intervention: active prophilactic barrier against skin breakdown
  Interventions: Device: Skin protective dressing device
- polyurethane film (Tegaderm) (Active Comparator): The polyurethane film is applied ss skin protective dressing device before NIV and kept on site till the 7th day of treatment Intervention: active prophilactic barrier against skin breakdown
  Interventions: Device: Skin protective dressing device
- Hydrocolloid (Duoderm) (Active Comparator): Hydrocolloid is applied ss skin protective dressing device before NIV and kept on site till the 7th day of treatment Intervention: active prophilactic barrier against skin breakdown
  Interventions: Device: Skin protective dressing device
- Control (No Intervention): In this no-intervention arm, any skin protective dressing devices is applied before NIV starting

INTERVENTIONS:
Device: Skin protective dressing device — Application of one the three indicated devices (3 active arms) to prevent NIV-induced skin injury
  Arms: Hydrocolloid (Duoderm); polyurethane film (Tegaderm); polyurethane foam (Allewyn adesive)

SUMMARY:
In patients with acute respiratory failure (ARF) undergoing noninvasive ventilation (NIV), the main complication of the use of the mask is the development of decubitus, sometimes so severe and painful as to force a suspension of the NIV itself . The lesions are mainly located at the nasal bridge, as at this level the skin thin and placed directly on the bone is particularly vulnerable to the injury as consequence of the friction and pressure induced by the movement of the mask. The strategy of prevention and treatment commonly adopted is the application of hydrocolloids.

However, precise data are lacking about the demonstration of the effectiveness of these devices and the possibility of using other protective devices.

The purpose of this study was to evaluate the usefulness of large-scale three different systems of protection vs. no protection in preventing the development of decubitus lesions in patients receiving NIV for an episode of ARF.

DETAILED DESCRIPTION:
NIV is a form of ventilatory support which is popular overall in the world. The patient interface most commonly used in the course of NIV is by far the nasal or oronasal mask. The main complication of the use of the mask is the development of decubitus, sometimes so severe and painful as to force a suspension of NIV. The decubitus is mainly located at the nasal bridge, as at this level the skin thin and placed directly on the bone. According to Meduri et al.(Chest 1996) the duration of NIV, age, type of respiratory failure, the pressure used for ventilation and the level of albumin did not influence the development of necrosis.

Severe skin injury with ulceration and necrosis occurs in approximately 10% of patients receiving NIV trained in services. In the multicenter evaluation of a new face mask dedicated to the NIV (Gregoretti et al, Intens Care Med 2002) describes the development of NIV-induced decubitus in 100% of the control group treated with masks "traditional", with an average grade of 2.79 on a scale of Assessment Standard ranging from 1 (erythema) to 4 (necrosis).

The strategy of prevention and treatment commonly adopted is the application of appropriately shaped hydrocolloids. However, the data relating to the use of protective systems for the prevention of NIV-induced decubitus are limited and controversial. In a first pilot study (Callaghan et al,Professional Nurse 1998, the authors compared the protective efficacy of two types of "dressing" (Granuflex, Spenco Dermal and 10 patients, 10 patients) vs a non-randomized control group (10 patients): 30 patients in total . In this work, which presents a problem of inter-observer variability, the "Granuflex group" (or Duoderm) showed a greater protective effect (3 vs. 7 lesions in "Spenco Dermal group" vs 9 lesions in the control group). Recently, in a larger study, Weng (Intensive Crit Care Nurs 2008) compared the efficacy of two devices (Tegaderm and tegasorb) vs. a control group in 90 patients (30 per group) undergoing NIV. The rate of lesions was significantly lower in the treated groups (53% Tegaderm; Tegasorb 40%) than in the control group (96.7%), with no significant difference between the two interventional arms on both the incidence and the timing of onset of injury.

Therefore, given the limited data currently available regarding both the effectiveness and the choice of a protective device and in consideration of the continuous expansion of NIV in the acute setting, in our opinion it's seems to us justified to perform a controlled study comparing different types of devices in terms of skin protection during NIV.

ELIGIBILITY:
Inclusion Criteria:

* Hypoxemic-hypercapnic acute respiratory failure (while in O2-therapy):

  1. pH<7.30,
  2. PaCO2>50 mmHg,
  3. PaO2/FiO2<250,
  4. respiratory rate>25/min and use of accessory respiratory muscles
* Pure Hypoxemic acute respiratory failure(while in O2-therapy):

  1. pH>7.35
  2. PaCO2< 50 mmHg
  3. PaO2/FiO2<250
  4. respiratory rate>25/min and use of accessory respiratory muscles

For both types of acute respiratory failure: Signed informed consent by the patient or next keen. Age more than 20 year's old

Exclusion Criteria:

1. cardiac arrest
2. severe hemodynamic instability (> 1 vasoactive amine for more than 24 hours)
3. acute coronary syndrome (instable angina/AMI)
4. refusal of NIV
5. anatomic abnormalities interfering with mask fitting
6. pre-existent nasal lesions;
7. NIV for< 24 hours
8. kwon hypersensitivity to hydrocolloid and polyurethane
9. cancel of informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-05 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Failure rate of the prevention of the facial mask ventilation-induced skin damage in the three interventional groups and in the control group | 7 days

SECONDARY OUTCOMES:
Mask-induced discomfort | 7 days
  Discomfort/pain consequent to NIV-induced skin damage with the different protective devices
Costs for skin protection | 7 days
  Amounts of costs due to prevention of NIV-induced skin damage with the different protective devices
Prediction of NIV-induced skin damage | 7 days
  Identification of the variables independently associated with the development of skin injury due to mask ventilation
Success of NIV | Up to 30 days
  Rate of success of NIV to avoid endotracheal intubation and death

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Scala, MD, FCCP, Study Chair — PULMONARY DIVISION WITH RESPIRATORY INTENSIVE CARE UNIT, S. DONATO HOSPITAL, AREZZO, ITALY
Locations (1):
- Pulmonary Division With Respiratory Intensive Care Unit, S. Donato Hospital, Arezzo, Italy, Lucca, Italy

REFERENCES:
- [Result] Weng MH. The effect of protective treatment in reducing pressure ulcers for non-invasive ventilation patients. Intensive Crit Care Nurs. 2008 Oct;24(5):295-9. doi: 10.1016/j.iccn.2007.11.005. Epub 2008 Feb 1. PMID 18242994